CLINICAL TRIAL: NCT00223847
Title: An Investigation of Constraint Induced Language Therapy for Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Maher, Lynn - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3091R
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia rehabilitation; Aphasia therapy; Constraint therapy; Language therapy
MeSH Terms: conditions — Aphasia; Stroke

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: Constraint Induced Language Therapy

INTERVENTIONS:
Behavioral: Constraint Induced Language Therapy

SUMMARY:
The purpose of this study is to investigate the effects of intensive, constraint induced language therapy (CILT) for individuals with chronic aphasia compared with traditional aphasia therapy. The specific objectives of the proposed research are to determine the effects of therapy type (CILT vs. traditional) and dose density (intensive or distributed) on speech therapy outcome. In addition, we will investigate the functional and qualitative impact of these interventions on functional communication.

DETAILED DESCRIPTION:
Objectives: Aphasia is an acquired language disorder that is a common sequelae of stroke and poses tremendous levels of handicap for the victim as well as burden for caregivers. While the efficacy of aphasia rehabilitation has been found to be statistically significant in its effect (Wertz et al., 1986; Robey, 1994), its clinical significance has been often disappointing (Siegel, 1987). A promising avenue for rehabilitation of chronic aphasia based on the approach and principles of Constraint Induced Movement Therapy (CIMT) has recently been described (Pulvermuller et al., 2001). These investigators reported that individuals with chronic, stable aphasia benefited (statistically as well as clinically) from language therapy designed to include attributes of CIMT (forced-use delivered in high doses over a relatively short period of time). In a limitation of the study, the conditions of constraint-induced language treatment (CILT) and traditional treatment were confounded by differences in treatment intensity. A pilot study funded by the VA Rehabilitation Research & Development (RR&D) to begin to control for confounding variables and treatment intensity is currently underway in a collaboration between the Houston VAMC Center of Excellence in Healthy Aging with Disabilities and the Brain Rehabilitation Research Center of Excellence in Gainesville, FL. While data collection is ongoing, preliminary results suggest that individuals with chronic aphasia made substantial, measurable change on a language battery following intensive CILT.

The purpose of this study is to expand on the pilot work we have done and to identify the functional and qualitative impact of these interventions on communication in naturalistic settings and on caregivers. Specifically, we will compare the relative impact of therapy type (constrained, forced speech TX vs. multi-modal PACE TX) and dose intensity (massed practice or distributed) on rehabilitation of chronic aphasia.

Research Plan: Using between group comparisons and multiple-baseline single subject comparisons, we will examine the impact of CILT in a larger group of individuals with aphasia, controlling for the confounding variables of massed practice, forced use and relevant context. In addition, we will investigate the functional and qualitative impact of these interventions on communication in naturalistic settings.

Methods: A total of 48 subjects collected at three sites (Houston, Gainesville and Tampa VAMCs) will be randomly assigned across four experimental conditions: 1) intensive CILT; 2) intensive PACE therapy; 3) distributed CILT and 4) distributed PACE therapy. Pre and post treatment language assessments, discourse samples, daily probe measures and qualitative interviews will be used to measure TX effects. In addition, these measures will be recollected one month following TX to assess the stability of the TX effects.

ELIGIBILITY:
Inclusion Criteria:

Moderate to moderately severe, non-fluent aphasia Unilateral Left CVA Right-handed Primary Language is English Adequate hearing and vision to participate in group therapy

Exclusion Criteria:

Multiple strokes HX of other neurological impairment (e.g. dementia) Non-English speaking Poor auditory comprehension Severe apraxia of speech

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Maher, PhD CCC/SLP, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States